CLINICAL TRIAL: NCT02574936
Title: Effects of Reduction Dead Space Volume With Karydakis Modification
Brief Title: Reduction Dead Space Volume With Karydakis Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siverek Devlet Hastanesi (Other)
Collaborators: Harran University (Other)
Responsible Party: Principal Investigator, Abdulcabbar Kartal, Principal Investigator, Siverek Devlet Hastanesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74059997.050.01.04/77
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: PILONIDAL SINUS
Keywords: karydakis modification; pilonidal sinus; complication
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- modified Karydakis,surgical technique (Other): a new surgical technique(modified Karydakis) to be compared with standard Karydakis
  Interventions: Procedure: A new surgical technique

INTERVENTIONS:
Procedure: A new surgical technique — Description of a new surgical technique in pilonidal sinüs surgery in order to reduce dead space volume.
  A flap extending across the cut (Karydakis) is prepared in medial edge of the wound, 1 cm deep and 2 to 3 cm to be towards the interior. Prepared flap is shifted to the medial and sutured to presacral fascia with vicryl 2/0. To reduce the volume of the dead space formed in the lateral, 5 mm skin is excised along the incision in the flap side. Skin is approximated with sutures in the form of intermittent, using 2/0 poliprolen. No drain used
  Other Names: Modified Karydakis

SUMMARY:
The purpose of this study is to reduce the volume of dead space by a modification in kardakis flap procedure and consequently, to reduce the use of drains, wound drainage, seroma and hematoma formation, skin degradation and recurrence rates.

DETAILED DESCRIPTION:
The study was a pilot study of 80 patients. Excluding criteria were previous sinüs surgery, active infection, patients who did not accept the procedure and patients under age of 18. After excision of the sinüs volume was measured using a beaker. A flap extending across the cut (Karydakis) was prepared in medial edge of the wound, 1 cm deep and 2 to 3 cm to be towards the interior. Prepared flap was shifted to the medial and sutured to presacral fascia with vicryl 2/0. To reduce the volume of the dead space formed in the lateral, 5 mm skin was excised along the incision in the flap side. Skin was approximated with sutures in the form of intermittent, using 2/0 poliprolen. No drain used. All patients were discharged on postoperative day 1. Sutures were removed 2 weeks later. All patients for at least 6 months were followed for wound drainage, seroma and hematoma formation, separation of skin and and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* patients who accept the procedure
* chronic p.sinüs disease

Exclusion Criteria:

* previous sinüs surgery
* active infection
* patients who did not accept the procedure
* patients under age of 18.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Effects of reducing the dead space volume (Change in dead space volume) with a modification in The Karydakis Method in sacrococcygeal pilonidal sinus surgery | 18 months
  OUTCOME MEASURE:
  1. Extracted sinus volume
  2. The number of patients with complications
     1. Delayed wound healing
     2. seroma
     3. hematoma formation
     4. wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Ali Uzunköy, Study Director — Harran University